CLINICAL TRIAL: NCT00082706
Title: Phase II Trial of 5-FU, Leucovorin, Gemcitabine, and Cisplatin for Adenocarcinomas of the Urothelial Tract and Urachal Remnant
Brief Title: Fluorouracil, Leucovorin, Gemcitabine, and Cisplatin in Treating Patients With Metastatic or Unresectable Adenocarcinoma of the Urothelium or Urachal Remnant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0111; P50CA091846 (NIH); ID-030111 (Other: UT MD Anderson Cancer Center); CDR0000355828 (Registry Identifier: NCI PDQ); NCI-2012-01305 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Urethral Cancer; Urachal Cancer
Keywords: adenocarcinoma of the bladder; recurrent bladder cancer; stage IV bladder cancer; recurrent urethral cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; stage III bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms; Urachal cancer | interventions — Fluorouracil; Leucovorin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5-FU, Leucovorin, Gemcitabine + Cisplatin (Experimental): 5-FU continuous infusion over Days 1 - 5; Leucovorin once a day as a short infusion on Days 1 - 5; Cisplatin infusion over a few hours (usually 2-4 hours) once a day on Days 1 - 5; Gemcitabine infusion over 30 minutes on Days 1 & 5 only.
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: 5-Fluorouracil (5-FU) — Day: 1 - 5 Dose: 200 mg/m2 IVCI daily x 5 days
  Other Names: 5-FU; Adrucil; Efudex
Drug: Leucovorin — Day: 1 - 5 Dose:10 mg/m2 daily x 5 days
  Other Names: Citrovorum; Wellcovorin
Drug: Cisplatin — Day: 1 - 5 Dose: 20 mg/m2 daily x 5 days
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Gemcitabine — Day: 1 & 5 Dose: 200 mg/m2 (Two doses only)
  Other Names: Gemcitabine Hydrochloride; Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, gemcitabine, and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving fluorouracil together with leucovorin, gemcitabine, and cisplatin works in treating patients with metastatic or unresectable adenocarcinoma of the urothelium or urachal remnant (part of the bladder).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate and overall survival of patients with metastatic or unresectable adenocarcinoma of the urothelium or urachal remnant treated with fluorouracil, leucovorin calcium, gemcitabine, and cisplatin.

Secondary

* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients are stratified according to diagnosis (adenocarcinoma of the urothelium vs adenocarcinoma of the urachal remnant).

Patients receive fluorouracil by vein (IV) continuously, leucovorin calcium IV once daily, and cisplatin IV once daily on days 1-5 and gemcitabine IV on days 1 and 5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3-6 months.

PROJECTED ACCRUAL: A total of 23-46 patients (7-18 with adenocarcinoma of the urachal remnant and 16-28 with adenocarcinoma of the urothelium) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proof of cancer originating from the urinary tract with adenocarcinoma as the predominant (>/= 50%) histology. Dr. Czerniak and/or Dr. Tamboli will be consulted in equivocal cases of mixed histology. The Study Chairman is the final arbiter in questions of mixed histology.
2. Bi-dimensionally measurable disease. All patients must have measurable or evaluable disease. In general, liver and lung lesions should be at least 1 cm, and patients with node-only disease should have lesions of >/= 1.5 cm in greatest dimension. Patients with disease confined to bone may be eligible if a measurable lytic defect, or soft-tissue component in present. Those without measurable disease may be eligible if a serum marker is elevated (>/= 4 x ULN) (ie: CEA, CA-125, CA19-9, bhCG, etc).
3. (# 2 cont'd) The Study Chairman is the final arbiter in questions related to measurability. Patients with a three-dimensional mass or pelvic sidewall fixation on bladder examination under anesthesia are considered to have measurable disease.
4. Patients are eligible if they have evidence of metastatic disease, or if their tumor is surgically unresectable. In the absence of grossly metastatic disease, all patients should be seen and evaluated by a member of the Urology staff to assess their potential for resection.
5. Patients must have adequate physiologic reserves as evidenced by: • Life expectancy of at least 9 months (based on co-morbidity) & at least 9 weeks based on the natural history of their cancer. • Zubrod Performance Status (PS) of </= 2; or 3 if of recent onset and due entirely to the cancer and not to comorbidity, and especially if the compromised performance status is due to uncontrolled pain which is expected to be rapidly reversible when therapy starts.
6. (#5 cont'd) • Adequate bone marrow function as defined by absolute neutrophil count >/= 1,800 and platelet count >/= 150,000. Supranormal values judged to be of benign or inconsequential etiology are acceptable. • Transaminase (either SGPT or SGOT) </= 2x the upper limit of normal. • Conjugated bilirubin </= 2x the upper limit of normal. • Creatinine clearance (either measured or estimated using the formula of Cockcroft and Gault) of >/= 35 mL/min: CLcr = [(140-age) • wt(kg)]/[72 •Creat (mg/dL)] (For females, x 0.85)
7. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of this hospital.
8. Patients must be at least 6 weeks out from pelvic irradiation, and must not have had more than 10% of the bone marrow irradiated.
9. Patients with a history of cardiac disease, or evidence of ischemic heart disease on EKG must have adequate cardiac function with an EF >/= 40% to participate.
10. Patient must be at least 18 years of age to participate in this study.

Exclusion Criteria:

1. Patients with metastases to the bladder from a primary adenocarcinoma arising outside the urinary tract are ineligible.
2. Overt psychosis or mental disability or otherwise incompetent to give informed consent.
3. A life threatening illness (unrelated to tumor) that would prevent completion of protocol therapy.
4. Pregnant or nursing women, as the drug therapy regimen, and support medications pose significant potential risks to the fetus and newborn.
5. Patients with second malignancies are eligible provided that the expected outcome from the second cancer is such that this will not interfere in the delivery of this therapy, or the assessment of response.
6. Patients with uncontrolled CNS metastases are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-04-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Response | Every 2 cycles (6 weeks)
  Complete Response: Participants counted as complete response if they have no radiological evidence of tumor, have no signs or symptoms of disease, and have normalized tumor markers (in those with initially elevated markers). Participants with an intact, tumor-containing bladder, must have a cystoscopy and exam under anesthesia to confirm a complete response. Partial response: Any response less than a complete response. Progressive disease: Progressive disease is at least 25% increase in tumor volume, or any new site of involvement, including the CNS. Increasing severity of symptoms, if judged by treating physician to be due to progressive disease, also counted as progression, even if these are not accompanied by an "objective" indicator. Any unequivocal increase (i.e. to greater than 5 mi.u./mL in beta-hCG) in a male patient taken to represent progressive disease, as will two consecutive rises amounting to a total of at least 125% of baseline for any other tumor marker.

SECONDARY OUTCOMES:
Number of Patients with Dose-Limiting Toxicity | Continous assessment during 21 day cycles
  For each single arm trial, a stopping boundary also imposed to monitor toxicity of the new combination chemotherapy. Trial should be stopped for the 90% probability that the dose-limiting toxicity is greater than 40%. Participants monitored in groups of 3 sequentially. Stopping boundary obtained using a Bayesian monitoring rule.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org